CLINICAL TRIAL: NCT01245998
Title: Prospective, Randomized, Double-blinded Trial of the Efficacy and Safety of Different Doses and Duration of Low Molecular Weight Heparin (Dalteparin) in Superficial Vein Thrombosis
Brief Title: Efficacy of Low Molecular Weight Heparin in Superficial Vein Thrombosis
Acronym: REVETR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Pavel POREDOS, professor tenure track, board certified in internal medicine, cardiology and vascular disease, head of the research department, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REVETR2010
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Superficial Thrombophlebitis
Keywords: Thrombophlebitis; Venous thrombosis; Pulmonary embolism; Anticoagulants; Low-Molecular-Weight Heparin
MeSH Terms: conditions — Thrombophlebitis; Venous Thrombosis; Pulmonary Embolism | interventions — Dalteparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dalteparin 5000 I.U./24 h s.c. (Active Comparator)
  Interventions: Drug: Dalteparin
- dalteparin 15000 I.U./24 h s.c. (Active Comparator)
  Interventions: Drug: Dalteparin

INTERVENTIONS:
Drug: Dalteparin — dalteparin 5000 I.U./24 h s.c. for 6 weeks
  Other Names: Fragmin
  Arms: dalteparin 5000 I.U./24 h s.c.
Drug: Dalteparin — dalteparin 15000 I.U./24 h s.c. for 6 weeks
  Other Names: Fragmin
  Arms: dalteparin 15000 I.U./24 h s.c.

SUMMARY:
The aim of the study is to establish whether treatment of superficial vein thrombosis (SVT) with low-molecular-weight heparin in preventive or therapeutic doses prevents disease progression and thromboembolic events (deep vein thrombosis and pulmonary embolism), whether efficacy of low-molecular-weight heparin differs with regard to the dosage used (prevention, treatment), and to recognize groups of patients in which treatment with heparin is most efficient, as well as to determine factors that influence the efficacy of SVT treatment with heparin.

DETAILED DESCRIPTION:
Until recently thrombophlebitis was regarded as a benign and self-limiting disease. Recent studies have shown that various complications, especially vein thrombosis and pulmonary thromboembolism, often accompany SVT. An observational study (Prospective Observational Superficial Thrombophlebitis - POST) showed that three months after onset of the disease thromboembolic events occurred in 10% of patients: pulmonary embolism in 0.4%, disease progression in 3.1% and disease recurrence in 1.9% of patients. Therefore, SVT is now frequently regarded as a part of the thromboembolic syndrome. On the basis of the evidence referred to above anticoagulants, especially heparin, are used more and more often for treatment of SVT instead of anti-inflammatory drugs and non-steroidal antirheumatics. Several studies performed so far have examined the efficacy of standard and low-molecular-weight heparin in various doses, but no final conclusion on the efficacy of treatment of SVT with heparin has been established yet.

A study by Marchiori and colleagues showed that 8-12-day treatment of SVT with preventive and therapeutic doses of low-molecular-weight heparin significantly reduces progression and relapse of the disease, but not its thromboembolic complications. Another study demonstrated that low-molecular-weight heparin in combination with elastic compression was not significantly more effective than compression alone. Comparison of preventive and therapeutic doses of low-molecular-weight heparin given to patients over the period of one month after disease onset showed no differences in the efficacy in prevention of disease progression and thromboembolic complications. The standard (unfractionated) heparin was also shown to be effective in preventing disease progression, however, but not in preventing thromboembolic complications. It is also not clear how long the treatment with heparin should last. So far only one study compared the efficacy of treatment with various doses of low-molecular-weight heparin from one month to three months' duration; it demonstrated that 1-month treatment with lower doses of heparin was as effective as 3-month treatment with therapeutic doses of heparin. A recent study (CALISTO) compared the efficacy of preventive doses of fondaparinux (2.5 mg) with placebo in more than 3,000 patients with SVT and concluded that anticoagulant treatment of SVT probably does not significantly influence prevention of thromboembolic complications (Abstract presented at the 5th Annual Meeting of the American Society of Hematology).

Results of recent studies show that heparin (standard or low-molecular-weight heparin) in various doses prevents SVT progression, but no final agreement has emerged as to whether they prevent the occurrence of thromboembolic complications. Interpretation of the results is difficult because of the heterogeneity of the patients included in certain studies and especially because of unavailability of subgroup analyses, which would help to establish whether treatment with heparin is more effective in certain groups of patients with SVT than in those with presenting forms of the disease. Latest (2008) guidelines for prevention of venous thromboembolic events adopted by the American College of Chest Physicians (ACCP) recommend treatment with at least preventive or median doses of low-molecular-weight heparin or standard heparin for the duration of not less than 4 weeks. This recommendation was based on a very low evidence level (level 2B).

In this study, we aim to investigate whether the extensiveness of thrombophlebitis and the proximal distance of the end of a blood clot from saphenofemoral and saphenopopliteal junction influence the efficacy of SVT treatment with heparin. The investigators shall also monitor the expression of systemic inflammatory parameters that might be related to the efficacy of the treatment and progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent to participate in the study
* symptomatic thrombophlebitis of the great saphenous vein measuring at least 10 cm or the small saphenous vein measuring at least 10 cm or a collateral of the great saphenous vein measuring at least 10 cm (within 7 days from the onset of the disease)
* age 18 to 85 years
* body weight 65 to 85 kg

Exclusion Criteria:

* inability to objectively confirm the diagnosis
* excessive or insufficient body weight (more than 85 kg or less than 60 kg)
* history of previous thromboembolic complications (including previous thrombophlebitis, vein thrombosis and pulmonary embolism)
* contraindications for anticoagulant treatment
* active bleeding or high risk for bleeding contraindicating treatment with (LMWH)
* diseases requiring anticoagulant treatment
* proximal or distal deep vein thrombosis or pulmonary embolism (either symptomatic or incidentally found asymptomatic)
* thrombophlebitis of the great saphenous vein at a distance of less than 5 cm from the saphenofemoral junction or thrombophlebitis of small saphenous vein at a distance of less than 3 cm from the saphenopopliteal junction
* thrombophlebitis that might arise as a consequence of a previous intravenous access (infusion thrombophlebitis), sclerotherapy or surgical treatment of chronic vein insufficiency
* pregnancy, known malignant disease or chemotherapy
* immobility
* advanced stage of kidney failure (GF < 30 mL/min/1.72 m2)
* significant liver disease (e.g., acute hepatitis, chronic active hepatitis, cirrhosis) or alanine transaminase (ALT) >\= 2 times the upper limit of normal (ULN), or total bilirubin (TBL) x 1.5 times the ULN

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2012-12-03 (Actual); Study Completion 2014-01-01 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and safety of low-molecular-weight heparin - dalteparin in patients with ST | 3 months
  To compare the efficacy of therapeutic vs. preventive doses of dalteparin in prevention of thromboembolic complications and disease progression in patients with acute thrombophlebitis of lower extremities
Combined end-point: occurrence of symptomatic or asymptomatic deep vein thrombosis, symptomatic pulmonary embolism or ultrasonographic blood clot progression or relapse of ST | 3 months
Clinically relevant bleeding occurring | during treatment
  (i.e., major or clinically relevant non-major bleeding)

SECONDARY OUTCOMES:
To investigate the safety of ST treatment with preventive doses of dalteparin compared with therapeutic doses, death, bleeding, heparin-induced thrombocytopenia (HIT) | 3 months
To ascertain whether the extent or progression of ST is related to systemic inflammatory parameters | 12 months
To study a possible correlation between effectiveness of treatment of ST with preventive and therapeutic doses of dalteparin and severity of systemic inflammatory parameters. | 12 months
To determine whether the extension of anticoagulant treatment with the study drug for additional six weeks is more effective and safer | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Poredos, M.D., Ph.D., Principal Investigator — University Medical Centre Ljubljana, Department of Vascular Disease
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Result] Spirkoska A, Jezovnik MK, Poredos P. Time course and the recanalization rate of superficial vein thrombosis treated with low-molecular-weight heparin. Angiology. 2015 Apr;66(4):381-6. doi: 10.1177/0003319714533183. Epub 2014 May 7. PMID 24807875